CLINICAL TRIAL: NCT06625905
Title: Musculoskeletal Ultrasound to Assess Myofascial Trigger Points: Developing a Comprehensive Methodological Framework
Brief Title: Ultrasound Assessment of Myofascial Trigger Points
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Diego Lapuente Hernández, Predoctoral Researcher and Collaborating Professor, Universidad de Zaragoza
Other Study IDs: PI24/215; RAT 2024-131 (Other: University of Zaragoza)
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Myofascial Pain; Myofascial Trigger Points; Musculoskeletal Pain
Keywords: Ultrasonography; Myofascial trigger point; Image analysis; Manual palpation
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Myofascial/musculoskeletal pain group (active myofascial trigger points): This group comprises individuals who present with myofascial and/or musculoskeletal pain, with the presence of at least one myofascial trigger point (MTrP) classified as active. Active MTrPs are characterized by the following criteria: a palpable taut band within the muscle, a hypersensitive spot within the band, and the reproduction of the patient's pain upon palpation. The selection of participants for this group will focus on individuals exhibiting active MTrPs in gastrocnemius medialis muscle.
  Interventions: Diagnostic Test: Ultrasound imaging
- Control group (participants without pain, latent or no myofascial trigger points): The control group consists of individuals who do not present with any musculoskeletal pain or dysfunction. These participants may or may not exhibit latent MTrPs. Latent MTrPs are defined as palpable taut bands and hypersensitive spots within the muscle that do not reproduce the patient's pain but may cause discomfort when palpated. Participants in this group will be recruited based on their lack of musculoskeletal complaints.
  Interventions: Diagnostic Test: Ultrasound imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging — Both groups of participants-those with myofascial and/or musculoskeletal pain and those without musculoskeletal alterations-will undergo a standardized intervention focused on the application of vibratory stimuli, alongside real-time ultrasound imaging. Vibratory stimuli will be applied directly to the region of interest, specifically over the identified MTrP in participants with active myofascial pain. In participants without musculoskeletal alterations, the stimuli will be applied either over a latent MTrP or in a randomly selected area of the gastrocnemius medialis muscle, ensuring a consistent methodology across both groups. Simultaneously, real-time ultrasound imaging will be performed to capture detailed images of the muscle tissue during the application of vibratory stimuli. Imaging will be conducted in two planes (longitudinally and transversely).

SUMMARY:
Musculoskeletal pain represents a significant burden on individuals and the healthcare system in Spain, where 20% of adults experience pain, and 7% suffer from it daily. Myofascial pain syndrome (MPS), one of the most frequent causes of musculoskeletal pain, affects over 85% of the general population at some point. MPS is characterized by local or referred pain and the presence of myofascial trigger points (MTrPs). Despite advancements in diagnostic technologies, the evaluation of MTrPs still largely relies on manual palpation due to the absence of conclusive findings for their objective identification.

Ultrasound presents a promising alternative as a widely available, cost-effective, and non-invasive diagnostic tool for MTrPs. While prior studies on ultrasound for MTrP detection have shown variable sensitivity and specificity (ranging from 33% to 100%), no consensus has been reached on a standardized ultrasound methodology for reliable clinical use. The ability to accurately identify MTrPs through ultrasound could shift the current paradigm, facilitating earlier diagnosis and preventing the chronicity of musculoskeletal pain, thus improving patient care and reducing healthcare costs.

This study aims to evaluate ultrasound as a potential gold standard for MTrP diagnosis and characterization. By exploring optimal ultrasound modes (B-mode, Doppler), we aim to standardize a highly reliable inter-examiner diagnostic protocol that can be easily applied in clinical practice using accessible technology, such as portable wireless ultrasound devices. Specific objectives include: 1) developing ultrasound exploration protocols for MTrP detection; 2) evaluating vibration parameters for enhanced MTrP visualization; 3) characterizing MTrPs through ultrasound by analyzing size, shape, location, and echotextural features; and 4) validating proposed protocols by correlating them with manual palpation and clinical measures.

This research will contribute significantly to understanding MTrPs, providing innovative diagnostic tools and protocols that will improve the precision and effectiveness of musculoskeletal pain assessment. The findings may also have important clinical implications for MTrP-related conditions, enhancing patient care and quality of life.

DETAILED DESCRIPTION:
This exploratory study aims primarily to characterize myofascial trigger points (MTrPs) and identify the optimal ultrasound protocol for their real-time visualization. Participants will be subjected to vibratory stimuli applied to the MTrP location.

As a secondary objective, the study will explore variations in ultrasound imaging of muscles without MTrPs, comparing measurements taken within the same muscle between different subjects. The goal is to establish a reference point for defining the normal range of various muscle echotexture values in ultrasound images of healthy individuals. This analysis will include metrics such as mean echogenicity, coefficient of variation of echogenicity, co-occurrence, and run-length matrices, among others.

To achieve this, the study will recruit subjects without musculoskeletal disorders (with or without latent MTrPs) and those with myofascial/musculoskeletal pain (with at least one active MTrP). Ultrasound images of the gastrocnemius medialis muscle, which has been selected because of the prevalence of MTrPs and its accessibility for palpation and ultrasound, will be analyzed.

To identify MTrPs in the selected muscle, both in participants with and without pain, at least two of the following diagnostic criteria must be met: 1) a palpable taut band within the muscle; 2) the presence of a hypersensitive spot within the taut band; and 3) referred pain when the MTrP is compressed. Although we are aware of the risk of false negatives, for participants with pain, to differentiate an active MTrP from a latent one, an active MTrP must reproduce the patient's symptoms, as both active and latent MTrPs commonly exhibit a taut band and hypersensitive spot.

The analysis of the data extracted from this study aims to discern any distinguishing features that could contribute to developing a model capable of accurately identifying MTrPs. This will involve using machine learning techniques or statistical modeling.

Additionally, the study will incorporate an analysis of the diagnostic reliability and validation of MTrP exploration protocol in superficial muscles, leveraging the recruited sample. This analysis aims to validate the MTrP exploration protocol by evaluating diagnostic reliability between ultrasound and manual palpation. Manual palpation is currently the most widely accepted criterion for MTrP diagnosis. An expert physiotherapist specialized in myofascial pain will use manual palpation to diagnose MTrPs in gastrocnemius medialis muscle. Using a dermographic pen, the exact area of the MTrP, as well as a control area outside the MTrP and tight band within the same muscle, will be marked. If no MTrP is detected, a random area within the muscle of interest will be marked instead. In both cases, a cross will be drawn to ensure precision in ultrasound probe placement for both longitudinal and transverse sections. This dual evaluation approach, combining manual palpation and ultrasound, aims to provide a comprehensive and reliable assessment of MTrPs in superficial muscles. The results will further clarify the effectiveness and accuracy of the MTrP exploration protocol, offering essential insights for clinicians and researchers involved in myofascial pain diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* For participants with myofascial/musculoskeletal pain, there must be at least one active myofascial trigger point (MTrP) in the gastrocnemius medialis muscle.
* Participants without pain may or may not have latent MTrPs in the gastrocnemius medialis muscle.

Exclusion Criteria:

* Any systemic medical condition, progressive neurological disease, active rheumatic disease, severe cardiac condition, malignant neoplasm, infection or acute vascular problems, fibromyalgia, myopathy, radiculopathy, myelopathy or other neuromuscular diseases.
* History of severe trauma or surgery in the last 6 months.
* Use of pacemakers or electronic implants.
* Pregnancy status.
* Obvious cognitive impairment and difficulties in communication, comprehension or cooperation.
* Physiotherapeutic treatment of a MTrP of the gastrocnemius medialis muscle with an Invasive Physiotherapy procedure (dry needling or percutaneous electrolysis) in the last month.
* Delayed onset muscle pain ("stiffness") after very intense exertion.
* Current use of any therapy (especially pharmacological) and/or any other substance that may affect the autonomic nervous system.
* Commonly accepted contraindications for Invasive Physiotherapy procedures (unbearable fear of needles, epilepsy or convulsions, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population from which the study groups or cohorts will be selected consists of individuals recruited through a variety of outreach channels coordinated by the research team. Recruitment efforts will include the dissemination of informational leaflets via multiple communication platforms, such as the official Instagram account of the iHealthy research group (@ihealthyeu) and the newsletter of the University of Zaragoza. Additionally, potential participants will be invited through direct communication with clients of the Valdespartera Physiotherapy Clinic (Zaragoza, Spain). The recruitment process will also involve collaboration with healthcare professionals, including physiotherapists and physicians, from several key institutions, such as the Lozano Blesa University Clinical Hospital, Miguel Servet Hospital, and the Seminario Health Center (Zaragoza, Spain). These professionals will be encouraged to inform their patients about the study and invite them to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Echovariation | At a single 1 day time point
  Echovariation is the primary variable of interest in this study. It refers to the variability of pixel intensities within an ultrasound image and is calculated as the ratio of the standard deviation to the mean echogenicity (brightness) of the image. This metric allows for an assessment of the texture and homogeneity of the tissue, providing insight into potential abnormalities such as the presence of myofascial trigger points (MTrPs). Echovariation is a key indicator of muscle tissue´s structural integrity and is critical in differentiating between healthy and pathological regions. The evaluation of echovariation will be conducted on ultrasound images captured from gastrocnemius medialis muscle in both longitudinal and transverse planes.

SECONDARY OUTCOMES:
Muscle thickness | At a single 1 day time point
  Muscle thickness refers to the greatest distance between the superior and inferior edges of a muscle, measured in millimeters. This variable provides a morphometric analysis of muscle size and is particularly useful for identifying any changes in muscle structure related to the presence of MTrPs. Ultrasound images will be used to measure the muscle thickness at predefined anatomical landmarks in the gastrocnemius medialis muscle.
Mean echogenicity | At a single 1 day time point
  Mean echogenicity refers to the average brightness level of the pixels in the ultrasound image. It is a measure of tissue density and is influenced by the structural composition of the muscle. In this study, mean echogenicity will be quantified to assess the relative brightness of muscle tissue in participants, with a focus on identifying any deviations that may indicate the presence of MTrPs or other pathologies.
Myofascial trigger point area | At a single 1 day time point
  The area of myofascial trigger points (MTrPs) will be calculated from ultrasound images by delineating the boundary of each identified trigger point. This provides an additional dimension to the morphometric analysis and offers insight into the size and spatial distribution of the MTrPs within the muscle tissue. The area will be measured in square millimeters and compared across participants with and without active MTrPs.
Grey Level Run-Length Matrices (GLRLM) | At a single 1 day time point
  GLRLM calculates statistics based on the length of consecutive pixels that have the same grey level in an ultrasound image. This method identifies the homogeneity of pixel intensities over specific regions of the image, contributing to the understanding of the internal architecture of the muscle. The GLRLM analysis will focus on determining the presence of consistent grey-level patterns that may be indicative of structural alterations in the muscle tissue related to MTrPs.
Pressure Pain Threshold (PPT) | At a single 1 day time point
  Pressure pain threshold (PPT) will be measured using a handheld pressure algometer, which quantifies the amount of pressure applied to a specific point on the body until the participant perceives pain. The measurement will be conducted with participants lying in a supine or prone position, depending on the muscle group being assessed. Three consecutive trials will be performed at 30-second intervals, and the mean value will be used for analysis, reported in kg/cm². Prior to measurement, participants will be familiarized with the algometer to ensure they can accurately identify when the sensation of pressure transitions into pain. The reliability of PPT measurements has been shown to be excellent when performed in triplicate within the same session.
Grey Level Co-occurrence Matrices (GLCM) | At a single 1 day time point
  GLCM is a texture analysis method used to quantify the spatial relationship between pairs of pixels within an ultrasound image. It measures the frequency and correlation of grey-level values at specific distances and angles within the image. This analysis will be performed on regions of interest in both healthy and pathological muscle tissue to asses tissue texture complexity and heterogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero Gallego, Principal Investigator — Universidad de Zaragoza; Eva María Gómez Trullén, Study Director — Universidad de Zaragoza
Locations (2):
- Spain (2):
  - Centro de Salud Romareda-Seminario, Zaragoza, Aragon
  - Faculty of Health Sciences of the University of Zaragoza, Zaragoza, Aragon

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: SAP, ICF
Time Frame: Once research has been published